CLINICAL TRIAL: NCT01134198
Title: Investigation of the Effects of Mifepristone (RU486) on Stress Sensitivity and Relapse Prevention in Cocaine Dependent Patients
Brief Title: Investigation of Mifepristone (RU486) on Stress Sensitivity and Relapse Prevention in Cocaine Dependent Patients
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Principal Investigator, Wilfrid Raby, Principal Investigator, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 6013; RU486 for Cocaine Dependence (Other Grant/Funding Number: NIDA K23 DA027044-01)
Record Dates: First submitted 2010-05-26; First posted 2010-05-31 (Estimated); Results first posted 2018-08-24 (Actual); Last update posted 2018-12-20 (Actual); Status verified 2018-11

CONDITIONS: Cocaine Dependence
Keywords: Cocaine Dependence
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Mifepristone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mifepristone (Active Comparator): Mifepristone 600mg
  Interventions: Drug: Mifepristone
- placebo (Placebo Comparator): Placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Mifepristone — Mifepristone 600mg, 3x/wk for 4 weeks
  Other Names: RU486
  Arms: Mifepristone
Drug: placebo — placebo
  Arms: placebo

SUMMARY:
This research will evaluate the impact of blocking central and peripheral glucocorticoid receptors on stress sensitivity and the risk of relapse to cocaine use in treatment-seeking cocaine-dependent individuals. Mifepristone (RU-486) will be the glucocorticoid antagonist used.

DETAILED DESCRIPTION:
This study attempts to reduce relapse risk by blocking glucocorticoid receptors, and thus allow some of the changes in the brain caused by cocaine to redress themselves

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 60.
2. Male.
3. Meets DSM?IV criteria for current cocaine dependence and is seeking treatment.
4. Identifies life stress (work, interpersonal, financial, etc) as a trigger for cocaine use or reports uncontrollable craving to use of cocaine.
5. Displays at least one cocaine-positive urine toxicology during screening.
6. Uses cocaine at least 4/30 days in the past month, or reports episodic binges of large amounts of cocaine (at least $200) at least 2x/month.
7. Able to give informed consent and comply with study procedures.

Exclusion Criteria:

1. Meets DSM-IV criteria for major depression, bipolar disorder, schizophrenia or any psychotic disorder other than transient psychosis due to drug abuse. Substance Induced Mood Disorder with Hamilton Depression Scale score ³13 will be excluded.
2. History of seizures in the last 2 years, or history of seizures related to the substance (cocaine, alcohol, or benzodiazepine) that the patient continues to use.
3. History of allergic, dermatological, or adverse event to mifepristone
4. Chronic organic mental disorder, insufficient proficiency in English that would render an individual incapable of giving informed consent.
5. Significant current suicidal risks, history of significant suicidal behavior or any suicide attempt within the past year.
6. Unstable physical disorders, which might make participation hazardous such as hypertension (>140/90), WBC < 3.5, new diagnosis of hepatitis (patients with chronic mildly elevated transaminase levels (£2-3 X upper limit of normal will be considered acceptable if PT/PTT is normal), renal failure (creat > 2; BUN > 40), or diabetes (HbA1c > 7%), and low Hb (< 12g/dL) or low Hct (<36%).
7. Coronary vascular disease as indicated by history, or suspected by abnormal ECG or history of cardiac symptoms. Hx of cardiac symptoms (chest pain, chest pressure, shortness of breath, syncope) during cocaine use.
8. Cardiac conduction system disease as indicated by QRS duration of ³ 0.11 msec.
9. Currently meets DSM-IV criteria for another substance dependence or abuse disorder other than nicotine, alcohol, or cannabis. If alcohol dependent, must not be in need of detoxification. Heavy male drinkers (who consume greater than 5 standard alcoholic drink per day per NIAAA definition) will be excluded.
10. Presents with metabolic indicators of hypoadrenalism such as low serum sodium (<130 mEq/L), high serum potassium (>5.5 mEq/L), Na/K ratio < 30:1, low fasting blood sugar (<50 mg/dL), or high BUN (>20 mg/dL), or a previous history of Addison's disease or adrenal insufficiency, or the presence of low K (< 3.5 mEq/L). spot AM cortisol <5ug/dL, PM cortisol < 3 ug/dL
11. Participants who cannot comply with study procedures during the initial hospitalization phase.
12. Supplemental exclusion criteria for cold pressor test (CPT): history of frostbite, open cut or sore on foot to be immersed, history of Raynaud's phenomenon. During the testing, if sBP > 190 or dBP > 120, or HR > 160, the test will be interrupted. A second occurrence of these values will stop all further CPT.

13: Patients taking medications metabolized by cytochrome 3A4 (ex: erythromycin, protease inhibitors) or that inhibit this cytochrome; or consuming grapefruit juice.

14: Patients with an underlying hemorrhagic disorder and those on anti-coagulants. INR > 1.1, PT > 17 msecs, total plt <100x109/L.

15: Use of treatment agents that inhibit steroid biosynthesis by the adrenal cortex, such as metyrapone, ketoconazole, fluconazole, aminoglutethimide, or etomidate. Patients also requiring inhaled steroids.

16. Female

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2010-05; Primary Completion 2016-09 (Actual); Study Completion 2018-02-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wilfid N Raby, Md, PhD, Principal Investigator — NYSPI
Locations (1):
- STARS, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Data has been presented as an oral presentation at the annual meeting of the College on Drug Dependence in Palm Springs California on June 16th 2016. The data is presently being prepared for publication in a peer-reviewed publication.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: the data will be available by the end of 2018, and will be indefinitely
Access Criteria: there will be no access criteria required

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 58 participants signed consent and were enrolled into the trial. Only 32 entered the randomized phase of the study with only 29 being assigned to one of the treatment arms.
Period: Phase 1
Arm/Group | Mifepristone | Placebo
Started (randomized in phase 1, inpatient stay) | 16 | 13
Completed (started phase 2, outpatient treatment) | 9 | 11
Not Completed | 7 | 2
Period: Phase 2
Arm/Group | Mifepristone | Placebo
Started | 9 | 11
Completed (completed phase 2) | 9 | 7
Not Completed | 0 | 4

BASELINE CHARACTERISTICS:
Population: demographics for 29 participants who were randomized and started Phase 1
Groups:
- Mifepristone: demographics for 16 participants who were randomized and started Phase 1.
  Mifepristone 600mg, 3x/wk for 4 weeks.
- Placebo: demographics for 13 participants who were randomized and started Phase 1.
  Placebo 600mg, 3x/week for 4 weeks
- Total: Total of all reporting groups
Arm/Group | Mifepristone | Placebo | Total
Number analyzed (Participants) | 16 | 13 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 46 (8.3) | 46 (8.3) | 46 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 16 | 13 | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 5 | 10
  Not Hispanic or Latino | 11 | 8 | 19
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 5 | 12
  White | 3 | 2 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Relapse by Days 10 and 28
Description: assessed percent of sample with documented cocaine use by days 10 and 28 based on self reported use and urine toxicology. Those with documented use were considered to have relapsed.
Time Frame: assessed during 8 weeks of trial, but reported for days 10 and 28 of trial
Population: participants entering phase 2 of trial
Measure: Count of Participants; unit: Participants
Arm/Group | Mifepristone | Placebo
Number analyzed (Participants) | 9 | 11
Participants
  Day 10: relapsed | 3 | 8
  Day 10: abstinent | 6 | 3
  Day 28: relapsed | 5 | 8
  Day 28: abstinent | 4 | 3

ADVERSE EVENTS:
Time Frame: Over 9 weeks (1 week of inpatient in phase 1 and 8 weeks in outpatient phase 2)
Arm/Group | Mifepristone | Placebo
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/13
Other Adverse Events (participants affected / at risk) | 13/16 | 5/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mifepristone (N=16) | Placebo (N=13)
nausea (Gastrointestinal disorders) | 5 (5) | 3 (3)
fatigue (General disorders) | 2 (2) | 1 (1)
constipation (Gastrointestinal disorders) | 2 (2) | 1 (1)
weakness (General disorders) | 2 (2) | 1 (1)
insomnia/hypersomnia (General disorders) | 2 (2) | 1 (1)
elevated eosinophils (Blood and lymphatic system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes